CLINICAL TRIAL: NCT06044714
Title: Effects of Acupuncture on Perceived Stress and Health in Military Service Members and Veterans
Brief Title: Effects of Acupuncture on Perceived Stress and Health in Military Service Members
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Collaborators: TriService Nursing Research Program (Other); University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Jane J. Abanes, Principal Investigator, United States Naval Medical Center, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMCSD.2022.0054
Record Dates: First submitted 2023-09-08; First posted 2023-09-21 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2025-05

CONDITIONS: Perceived Stress
MeSH Terms: interventions — Mindfulness-Based Stress Reduction

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual Standardized Stress Acupuncture (MSSA) and Mindfulness-Based Stress Reduction (MBSR) (Experimental)
  Interventions: Procedure: Manual Standardized Stress Acupuncture (MSSA); Behavioral: Mindfulness-Based Stress Reduction (MBSR)
- Mindfulness-Based Stress Reduction (MBSR) (Active Comparator)
  Interventions: Behavioral: Mindfulness-Based Stress Reduction (MBSR)

INTERVENTIONS:
Procedure: Manual Standardized Stress Acupuncture (MSSA) — Participants in the experimental group will receive 4 weekly sessions of MSSA, which consists of 8 acupuncture points: bilateral auricular (ear) shen men, GV- 20, GV-24.5 (Yin Tang), bilateral LI-4, and bilateral LR-3. Needles are left in situ for 30 minutes per session.
  Arms: Manual Standardized Stress Acupuncture (MSSA) and Mindfulness-Based Stress Reduction (MBSR)
Behavioral: Mindfulness-Based Stress Reduction (MBSR) — Participants will receive four sessions of MBSR group psychotherapy (no more than 10 participants per group session) via Microsoft Teams. The first session will be 90 minutes followed by three 60-minute weekly sessions.

SUMMARY:
The goal of this is to investigate the effect of a Manual Standardized Stress Acupuncture (MSSA) protocol as an adjunct treatment to a short-term mindfulness therapy for perceived stress and general health in service members (i.e., active duty military personnel and veterans).

The specific aims of this study are Aim 1) To evaluate the effectiveness of a brief MSSA as an adjunct treatment with a short-term Mindfulness-Based Stress Reduction (MBSR) compared with MBSR alone for perceived stress and general health in service members. Aim 2) To describe any perceived benefits of MSSA as an adjunct treatment with MBSR compared with MBSR alone for perceived stress and general health.

Participants will be asked to complete an informed consent if eligible for the study and randomized into two groups: 1) Participants in the experimental group will receive MSSA in addition to MBSR. 2) Participants in the control group will receive MBSR only. Researchers will compare experimental and control groups to see if the interventions mitigated perceived stress and improved the health of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Active duty and veteran service members,
* 18 to 65 years of age, self-report of perceived stress symptoms for at least one month,
* a score of 16 or above on the PSS,
* stable on psychiatric and other medications including blood pressure agents for at least three months,
* agrees to participate in group psychotherapy (i.e., MBSR), and
* able to provide informed consent.

Exclusion Criteria:

* Recent surgery within one month,
* alcohol abuse or dependence diagnosis within one month,
* active substance use/abuse/dependency treatment within one month,
* pregnant women (acupuncture can result in an induction of labor and spontaneous abortion on rare occasions), and
* has had acupuncture treatment, dry needling, and MBSR provided by a provider in the past month.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Perceived Stress Scale (PSS) | At baseline, at two weeks post interventions, and at four weeks post interventions
  The PSS is a 10-item scale used to evaluate perceived stress experience in adults. Perceived general stress is rated on a 5-point Likert-type scale ranging from never to very often. The total possible scores for PSS range from 0 to 56, with higher scores indicating higher stress.

SECONDARY OUTCOMES:
Insomnia Severity Index | At baseline, at two weeks post interventions, and at four weeks post interventions
  The ISI is a seven-item standardized self-report questionnaire that measures the subjective symptoms of insomnia. These subjective symptoms include the respondents' concerns and distress because of problems with sleep. The ISI measure contains seven items: perceived difficulty with sleep-onset, sleep maintenance, and early morning awakenings; satisfaction with sleep patterns; interference of sleep problems with daily functioning; impairment because of a sleep problem; and degree of distress or concern with the sleep problem. Each item in the ISI is rated from 0 to 4 whereby the higher number indicates more difficulty. The scores are added to yield a range of total scores from 0 to 28 in which a higher score suggests more severe insomnia.
The Short Form (SF) Health Survey | At baseline, at two weeks post interventions, and at four weeks post interventions
  The 20-Item Short Form Health Survey (SF-20) measures the multidimensional concept of health including perceptions about general health, physical health, mental health, and social functioning. Scores are transformed to a scale of 0 to 100 wherein high scores indicate better functioning.
Journal Log | At weeks 2 and 4 after treatments have been completed.
  Journal entries will include five open-ended questions about the participants' perceived benefits of treatment.

OTHER OUTCOMES:
Blood Pressure (systolic and diastolic) | Prior to each acupuncture session (experimental group only)
  Blood pressures will be measured using a vital signs measuring device
Heart Rate | Prior to each acupuncture session (experimental group only)
  Heart rate will be measured using a vital signs measuring device
Defense and Veterans Pain Rating Scale (DVPRS) | Prior to each acupuncture session and at the end of each acupuncture session (experimental group only)
  The DVPRS measures pain from 0 (no pain) to 10 (as bad as it could be)

CONTACTS AND LOCATIONS:
Locations (1):
- Naval Medical Center, San Diego, San Diego, California, United States